CLINICAL TRIAL: NCT02989259
Title: The Clinical Study of Apatinib for Patients With Advanced Non-squamous Head and Neck Cancer
Brief Title: Apatinib for Advanced Non-squamous Head and Neck Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Xiaohui He, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-H&N-008-1
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Head and Neck Neoplasms
Keywords: apatinib; advanced head and neck cancer; non-squamous
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- apatinib (Experimental): apatinib 500mg p.o. qd
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — apatinib 500mg p.o. qd
  Other Names: ApatinibMesylate tablet

SUMMARY:
In this study, the investigators try to evaluate the efficacy and safety of apatinib in advanced non-squamous head and neck cancer and to validate the correlative biomarkers.

DETAILED DESCRIPTION:
There is no standard therapy for patients with advanced (unresectable, locally advanced, recurrent or metastatic) non-squamous head and neck cancer. Apatinib is a novel vascular endothelial growth factor receptor 2 tyrosine kinase inhibitor, which has been approved for the treatment of patients with advanced gastric cancer refractory to two or more lines of prior chemotherapy. Vascular endothelial growth factor is highly expressed in non-squamous head and neck cancer and its expression correlates with stage, tumour size, vascular invasion, recurrence and metastasis. In this study, the investigators try to evaluate the efficacy and safety of apatinib in advanced non-squamous head and neck cancer and to validate the correlative biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 75 years;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2;
* Life expectancy of more than 12 weeks;
* At least one measurable lesion according to RECIST 1.1 which has not received radiotherapy =< 3 months;
* Histologically confirmed advanced (unresectable, locally advanced, recurrent or metastatic) non-squamous head and neck cancer, including adenocarcinoma, mucoepidermoid carcinoma, acinar cell carcinoma and adenoid cystic carcinoma;
* Recurrent and or metastatic lesions which are not suitable for local treatment;
* For patients with mucoepidermoid carcinoma, acinar cell carcinoma or adenoid cystic carcinoma, metastatic disease documented as having shown progression on a scan (CT, MRI) compared to a previous scan taken at any time in the past 12 months;
* For patients with adenocarcinoma, one regimen of prior chemotherapy was received for recurrent and or metastatic diseases;
* Adequate hepatic, renal, heart, and hematologic functions: absolute neutrophil count (ANC) ≥ 1.5×109/L, platelet count (PLT) ≥ 100×109/L, hemoglobin (HB) ≥ 90 g/L, total bilirubin (TBIL) ≤ 1.5×upper limit of normal (ULN), alternate aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 2.5×ULN (or ≤ 5×ULN in patients with liver metastases), Serum Cr ≤ 1×ULN, Cr clearance ≥ 50 mL/min, international normalized ratio (INR) < 1.5 or PT < ULN+4s or activated partial thromboplastin time (APTT) < 1.5×ULN, proteinuria < (++) or urinary protein ≤ 1.0 g/24 hrs;
* For women of child-bearing age, the pregnancy test results (serum or urine) within 7 days before enrolment must be negative. They will take appropriate methods for contraception during the study until the 8th week post the last administration of study drug. For men (previous surgical sterilization accepted), will take appropriate methods for contraception during the study until the 8th week post the last administration of study drug.
* Signed informed consent.

Exclusion Criteria:

* Accumulation of coelomic fluid (e.g. pleural effusion, ascites fluid, cardiac effusion) requiring treatment;
* Other malignancy within the past five years other than basal cell skin cancer, or carcinoma in situ of the cervix;
* Factors affecting the oral medication (e.g. inability to swallow, chronic diarrhea and intestinal obstruction);
* Major injuries and/or surgery =< 4 weeks prior to registration with incomplete wound healing. Patients who have received radiotherapy (except local palliative radiotherapy), chemotherapy, molecular targeted therapy =< 3 weeks, or nitrosoureas/mitomycin chemotherapy =< 6 weeks prior to registration;
* Patients with poor-controlled arterial hypertension (systolic pressure ≥ 140 mmHg and/or diastolic pressure ≥ 90 mm Hg) despite standard medical management;
* Suffered from grade II or above myocardial ischemia or myocardial infarction, uncontrolled arrhythmias (including QT interval male ≥ 450 ms, female ≥ 470 ms). Grade III-IV cardiac insufficiency according to New York Heart Association (NYHA) criteria or echocardiography check: left ventricular ejection fraction (LVEF)<50%;
* History of clinically significant haemoptysis =< 2 months (more than half of one tea spoon of fresh blood per day) prior to registration. Coagulation disfunction, hemorrhagic tendency or receiving anticoagulant therapy;
* History of clinically relevant major bleeding event (e.g. gastrointestinal hemorrhage, bleeding ulcer, occult blood ≥ (++), and vasculitis) =< 3 months prior to randomization;
* Patients who have active brain metastases or leptomeningeal disease. Patients with treated brain metastases are eligible if they are clinically stable with regard to neurologic function, off steroids after cranial irradiation ending at least 3 weeks prior to randomization, or after surgical resection performed at least 3 weeks prior to randomization. No evidence of Grade greater than or equal to 1 central nervous system (CNS) hemorrhage based on pretreatment CT or MRI scan;
* Centrally located tumors of local invasion of major blood vessels, or distinct interstitial lung disease by the chest radiographic findings (CT or MRI);
* Treatment with other investigational drugs or other anti-cancer therapy;
* Previous therapy with other VEGFR inhibitors (other than bevacizumab);
* Treatment in another investigational trial =< 4 weeks prior to registration;
* History of hypersensitivity to apatinib and/or the excipients of the trial drugs;
* Active or chronic hepatitis C and/or B infection, or other active uncontrolled infection;
* History of immunodeficiency disease (including HIV positive), concurrent acquired or congenital immunodeficiency syndrome, or history of organ transplantation;
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess =< 6 months prior to registration;
* History of arterial or venous thromboembolic events (e.g. cerebrovascular accident, cardiovascular accident, deep venous thrombosis and pulmonary embolism) =< 12 months prior to randomization;
* Administration of strong/potent cytochrome P450 (CYP)3A4 inhibitors within 7 days, or inducers within 12 days;
* Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study;
* History of mental diseases;
* Other conditions regimented at investigators' discretion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Response Rate | up to 3 years

SECONDARY OUTCOMES:
Progression-free survival | up to 3 years

OTHER OUTCOMES:
Overall survival | up to 3 years
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 3 years
serum soluble VEGFR2 | baseline
tumor phosphorylated VEGFR2 (p-VEGFR2) expressions | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui He, B.D., Principal Investigator — Cancer Hospital, Chinese Academy of Medical Sciences (CAMS) & Peking Union Medical College (PUMC)
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences (CAMS) & Peking Union Medical College (PUMC), Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li J, Qin S, Xu J, Xiong J, Wu C, Bai Y, Liu W, Tong J, Liu Y, Xu R, Wang Z, Wang Q, Ouyang X, Yang Y, Ba Y, Liang J, Lin X, Luo D, Zheng R, Wang X, Sun G, Wang L, Zheng L, Guo H, Wu J, Xu N, Yang J, Zhang H, Cheng Y, Wang N, Chen L, Fan Z, Sun P, Yu H. Randomized, Double-Blind, Placebo-Controlled Phase III Trial of Apatinib in Patients With Chemotherapy-Refractory Advanced or Metastatic Adenocarcinoma of the Stomach or Gastroesophageal Junction. J Clin Oncol. 2016 May 1;34(13):1448-54. doi: 10.1200/JCO.2015.63.5995. Epub 2016 Feb 16. PMID 26884585
- [Result] Le Tourneau C, Razak AR, Levy C, Calugaru V, Galatoire O, Dendale R, Desjardins L, Gan HK. Role of chemotherapy and molecularly targeted agents in the treatment of adenoid cystic carcinoma of the lacrimal gland. Br J Ophthalmol. 2011 Nov;95(11):1483-9. doi: 10.1136/bjo.2010.192351. Epub 2010 Dec 22. PMID 21183517